CLINICAL TRIAL: NCT03410407
Title: Central Nervous System (CNS) Involvement in Acute Myeloid Leukemia (AML): an Observational Retrospective Multicentre Study on Patients Previously Registered in GIMEMA Clinical Trials
Brief Title: Central Nervous System (CNS) Involvement in Acute Myeloid Leukemia (AML)
Acronym: AML1617
Status: Terminated | Type: Observational
Why Stopped: lack of interest
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML1617
Record Dates: First submitted 2018-01-11; First posted 2018-01-25 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Central Nervous System; Relapse; Prognostic factors
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML patients: AML patients according to the French-American-British (FAB) criteria, previously enrolled in GIMEMA Studies for AML treatment. AML patients with CNS involvement defined by the confirmation of leukemic blast cells in the centrifuged cerebrospinal fluid (CSF) with the presence of more than five WBCs in the CSF or the detection of a CNS granulocytic sarcoma using computed tomography or magnetic resonance imaging.
  Interventions: Other: Observation of CNS involvement

INTERVENTIONS:
Other: Observation of CNS involvement — AML patients with CNS involvement defined by the confirmation of leukemic blast cells in the centrifuged cerebrospinal fluid (CSF) with the presence of more than five WBCs in the CSF or the detection of a CNS granulocytic sarcoma using computed tomography or magnetic resonance imaging.

SUMMARY:
The present study aims at evaluating the prognostic factors at diagnosis predicting Central Nervous System (CNS) relapse in order to identify a group of patients with higher risk of CNS involvement in which prophylaxis with liposomal Ara-C or other drugs should be indicated.

DETAILED DESCRIPTION:
CNS involvement in AML is a rare event, poorly detailed in literature. Few data are available in pediatric cases, and less frequent in adult cases. Predisposing factors for AML adult patients with CNS involvement include young age, higher level of lactate dehydrogenase and white blood cells (WBC) counts at diagnosis, FAB M4 and M5 morphology, chromosome 16 inversion and chromosome 11 abnormality. No consensus exists regarding the treatment of AML patients with CNS involvement. Protocols used for AML treatment are largely based on high doses of cytarabine, which penetrate the blood brain barrier. On the contrary of acute lymphoid leukemia (ALL), prophylaxis with intrathecal chemotherapy is not routinely used in AML. Roudoski et al. showed that, when lumbar puncture (LP) was performed in 1,370 patients, only if clinically indicated, CNS disease was detected in 45 (3.3%) patients. Another 42 patients underwent routine LP as part of an investigational protocol, and in 8 (19%) CNS disease was detected (P<0.0001). Risk factors included high LDH, African-American ethnicity, and young age. Patients receiving high-dose cytarabine and those that did not had similar rates of CNS involvement. Disease free survival (DFS) and overall survival were shorter in patients with CNS involvement. Treatment in case of CNS involvement is not well established; the potential acute and long-term complications associated with cranial irradiation often limit its use. Prognosis remains poor also with high doses of cytarabine and/or therapeutic intrathecal chemotherapy. Castagnola et al. reported showed the outcome of 9 patients woth CNS+ AML: NSL was treated as follows: 4 patients received combined systemic HD Ara-C, cranial radiation therapy and intrathecal (IT) methotrexate (MTX); a second group of 4 patients was treated with HD Ara-C, IT MTX without cranial irradiation; HD Ara-C alone was administered in one patient. All patients of the first group and 2 patients of the second who achieved a complete remission (CR) had a median survival of 10 months after CNS involvement, while for the non-remitters it was 2 months. The unique durable response was observed after allogeneic bone marrow transplantation. Sanders et al. reported that craniospinal irradiation with or without intrathecal chemotherapy appears to be effective at eliminating leukemia in the craniospinal axis. However, the eradication of disease in the CNS was not found to be effective at preventing disease recurrence in the bone marrow, and despite improved control of disease in the CNS, adult patients with a CNS recurrence still had a poor prognosis. Furthermore, the rapidly fatal course of disease prevented an assessment of the durability of CNS response to irradiation. Aoki et al reported that allogeneic haematopoietic stem cell transplantation (HSCT) might improve outcomes for CNS+AML and Bar et al, showed that presence of CNS pre-HCT had no independent influence on post transplant outcome, which was primarily influenced by status of systemic disease at time of HCT. Due to the rarity of the disease we want to collect the data about CNS involvement, either at diagnosis or along the course of the disease, in AML patients already registered in previous GIMEMA Studies, trying to identify incidence, prognosis, prognostic factors and the best adequate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws (if applicable).
* Patients aged ≥18 years affected by AML according to the FAB criteria, previously enrolled in GIMEMA Studies for AML treatment. AML patients with CNS involvement defined by the confirmation of leukemic blast cells in the centrifuged cerebrospinal fluid (CSF) with the presence of more than five WBCs in the CSF or the detection of a CNS granulocytic sarcoma using computed tomography or magnetic resonance imaging.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia (FAB M3 subtype), antecedent haematological diseases or therapy-related AML.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AML patients previously enrolled in GIMEMA studies for AML treatment
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Number of CNS relapses | At 12 months from study start
  To estimate the association between biological and clinical characteristic at diagnosis and the occurrence of CNS relapse and to confirm predisposing factors already described in literature (young age, higher level of lactate dehydrogenase; WBC counts at diagnosis, FAB M4 and M5 morphology, chromosome 16 inversion and chromosome 11 abnormality) in AML patients previously registered in GIMEMA Studies and treated according to the GIMEMA AML protocols

SECONDARY OUTCOMES:
Number of patients in complete response | At 12 months from study start
  Estimation of the association between presence of CNS involvement at diagnosis and during the course of the disease, in terms of CR rate, Overall Survival (OS) and Disease Free Survival (DFS).
Number of patients alive | At 12 months from study start
  Estimation of the association between presence of CNS involvement at diagnosis and during the course of the disease, in terms of CR rate, Overall Survival (OS) and Disease Free Survival (DFS).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pulsoni, Study Chair — Dipartimento di Biotecnologie Cellulari ed Ematologia, "Sapienza", Università di Roma; Livio Pagano, Study Director — Dipartimento di Biotecnologie Cellulari ed Ematologia, "Sapienza", Università di Roma
Locations (14):
- Italy (14):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Aou Maggiore Della Carita' Di Novara - Scdu Ematologia, Novara
  - Ao Di Perugia, Ospedale S. Maria Della Misericordia - Ematologia E Trapianto Midollo Osseo, Perugia
  - Asl Di Piacenza, Ospedale "Guglielmo Da Saliceto" - Ematologia E Centro Trapianti, Piacenza
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Dipartimento di Biotecnologie Cellulari ed Ematologia, "Sapienza", Università di Roma, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Asui Di Udine - Presidio Ospedaliero "Santa Maria Della Misericordia" - Clinica Ematologica, Udine